CLINICAL TRIAL: NCT05360758
Title: Ibrutinib Adapted to Response in Patients Diagnosed With Chronic Lymphatic Leukemia
Brief Title: Ibrutinib Adapted to Response in Patients With CLL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Responsible Party: Sponsor
Other Study IDs: GATLA 11-LLC-21
Record Dates: First submitted 2022-04-27; First posted 2022-05-04 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Ibrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with CLL with treatment criteria, first line or relapsed/refractory.
  Interventions: Other: Evaluation of response to treatment with response-tailored Ibrutinib in patients with chronic lymphocytic leukemia

INTERVENTIONS:
Other: Evaluation of response to treatment with response-tailored Ibrutinib in patients with chronic lymphocytic leukemia — Evaluation of response to treatment with response-tailored Ibrutinib in patients with chronic lymphocytic leukemia using laboratory tests, abdominal ultrasound, general condition of the patient and bone marrow

SUMMARY:
As everyone knows in clinical practice, Ibrutinib dose reduction in patients with CLL with good response does not alter disease-free survival (DFS) or increase the risk of transformation.

Supported by the evidence of retrospective studies that have shown parity in DFS and OS between a group with standard treatment and another in which the dose of ibrutinib was reduced and others in which no significant differences were observed in the saturation point of the BTK receptor with good clinical response, even comparing plasma and intracellular pharmacokinetics and BTK occupancy together with the pharmacodynamic response, we propose to carry out a prospective response-adapted study with the aim of potentially reducing the rate of adverse events and improving the cost/benefit ratio of this therapy. Evaluating the efficacy and safety of Ibrutinib dose appropriate to the response in patients diagnosed with CLL.

DETAILED DESCRIPTION:
Chronic lymphatic leukemia is the most common form of leukemia in adults, most often arising from a malignant clone of B cells with a characteristic phenotype. It is far from uniform in presentation and clinical course. About a third of patients never require treatment and have a long survival; in another third, an initial indolent phase is followed by disease progression; the remaining third of patients have aggressive disease at onset and require immediate treatment.

The development of the Rai and Binet staging systems has allowed the division of patients with chronic lymphocytic leukemia into three prognostic groups: good, intermediate and poor prognosis.

The two staging systems have improved the identification of patients who need immediate treatment.

In recent years, a variety of new kinase inhibitors have been designed that target various components of the BCR signaling pathway. Targets primarily include phosphatidylinositol 3'kinase (PI3K) and Bruton's tyrosine kinase (BTK). All of these new drugs share a response pattern that results in nodal reduction and increased lymphocytosis, reflecting modulation of the microenvironment, which could prevent these cells from receiving survival signals emitted by the microenvironment. More importantly, these drugs appear to be able to bypass p53 deletion, raising the possibility that they may target existing proliferative pools in the bone marrow and lymph nodes, thus bringing therapy closer to curing p53. disease.

The treatment of chronic lymphatic leukemia (CLL) represents the paradigm of advances in the therapy of hematological neoplasms. In its beginnings, CLL therapy used monodrugs that gradually led to their combination in duplets and triplets with which results never before obtained were achieved. The development of Ibrutinib was probably the milestone that marked the importance of the signaling pathways of leukemic cells in the progression of the disease, opening the investigation of new target drugs that constitute the basis of current treatment in CLL.

The treatment paradigm changes with the approval of BTK (Bruton tyrosine kinase) (iBTK) inhibitors in patients with del17p and/or TP53 (MTP53) mutations, which have achieved overall survival results that have never been achieved before. Quickly after the randomized study of the first-generation iBKT Ibrutinib (I) vs Cl (Resonate 2), this iBTK achieved approval for first-line treatment in all patients. Shortly thereafter, the second generation iBTK acalabrutinib (A) is approved. In June 2020, the National Cancer Center Net (NCCN) guidelines place these agents as preferred in the initial treatment of CLL and make them the agents of choice among North American experts.

According to the study by Mato based on 197 patients, parity in DFS and OS between one group and another has been shown when the ibrutinib dose is reduced. In more than half of the cases, the dose reduction was by medical decision even in the absence of adverse effects.

No significant differences in the saturation point of the BTK receptor with good clinical response with reduced dose are observed in a pharmacokinetic and pharmacodynamic study carried out by Advani et al.

Chen et al carried out a pilot study on 11 patients reducing the dose in 3 phases starting with the standard, a second phase with 280mg/day and a third at 140mg/day, comparing plasmatic and intracellular pharmacokinetics and the occupation of BTK together with the response pharmacodynamics, showing that the lowest dose was sufficient to occupy >95% of the BTK receptor and inhibit the downstream BTK signal.

Despite the improvements in outcomes for patients with poor-prognosis Chronic Lymphocytic Leukemia seen with ibrutinib, these patients are rarely cured. To further improve the results obtained, reduce the toxicity generated from prolonged treatment and reduce the costs of therapy, this protocol is proposed based on a dose adapted to the response to personalized treatment in each patient who meets the initial criteria. of treatment.

This is a prospective, open-label, multicenter, uncontrolled phase II study to evaluate the response to reduced doses of ibrutinib after achieving complete hematologic response or persistent partial response (for 3 or more months), in patients diagnosed with CLL with criteria treatment, first line or relapsed / refractory.

The study design consists of 2 phases:

PHASE I: Treatment with Ibrutinib 420mg/day (3 capsules). Laboratory controls, physical examination with cardiological evaluation will be performed every 14 days during the first 3 months, then every 3 months.

PHASE II: Upon achieving complete hematologic or sustained partial remission for more than 3 months, the Ibrutinib dose is reduced to 280 mg per day (2 capsules). Controls will be carried out every 2 months for 6 months. If complete/partial response is sustained, continue with checkups every 3 months.

Patients who reach phase II, at 6 months, CFM will be performed in peripheral blood. If MRD is negative, CFM should be performed on the bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CLL with criteria for starting treatment.
* Patients diagnosed with relapsed/refractory CLL.
* Patients diagnosed with CLL not exposed to iBTK.
* Patients with a diagnosis of CLL older than 18 years.
* Patients who have been diagnosed within the six months prior to the start of the registry will also be eligible, if they are followed prospectively by the participating centers and the required information is available.
* Signature of the informed consent.
* Patients who understand the risk of pregnancy during treatment and are willing to use safe contraceptive methods.

Exclusion Criteria:

* CLL without criteria for starting treatment.
* Small cell lymphocytic lymphoma.
* Previous exposure to iBTK.
* HIV positive, hepatitis B or C positive (unless there is vaccination), Chagas positive or HTLV-1 positive.
* Performance Status (ECOG) >= 3.
* Second active malignancy currently requiring treatment (with the exception of basal cell carcinoma).
* Class III or IV heart failure, previous acute myocardial infarction, unstable angina, ventricular tachyarrhythmias requiring treatment, severe COPD with hypoxemia, uncontrolled DBT or uncontrolled hypertension, active gastric ulcer.
* Active viral, bacterial, or fungal infection.
* Impaired renal function with clearance < 40 mL/min.
* BT/BD, GOT/GPT x 2.
* Mental deficiency that prevents adequate understanding of the treatment requirements.
* Thrombocytopenia (<30,000).
* Use of oral anticoagulants.
* Pregnancy / Lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with CLL with treatment criteria, first line or relapsed/refractory in Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate Progression Free Survival (PFS) in patients diagnosed with Chronic Lymphocytic Leukemia who undergo the treatment scheme protocolized by GATLA. | 24 months
Determine global response rate with dose reduction. | 24 months
Determine duration of response with dose reduction. | 24 months

SECONDARY OUTCOMES:
Evaluate Overall Survival (OS) in patients diagnosed with Chronic Lymphocytic Leukemia who undergo the treatment scheme protocolized by GATLA. | 24 months
Assess rate of adverse events grade 3 or more. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bertini, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda; Raimundo F Bezares, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda

IPD SHARING:
Plan to Share IPD: Yes
Share study protocol
Supporting Information: Study Protocol
Time Frame: The data will become available on June 2022, and will remain available until the end of the clinical trial.